CLINICAL TRIAL: NCT03965065
Title: Comparison of Sutureless Vs. Standard Biological Prostheses for Surgical Aortic Valve Replacement: a Randomised Multicenter Study (Madrid, Spain)
Brief Title: Comparison of Sutureless Vs. Standard Biological Prostheses for Surgical Aortic Valve Replacement
Acronym: COPERA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Manuel Carnero Alcazar, Adult Cardiac Surgeon, MD, PhD, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19/153-R_P
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Heart Valve Prosthesis; Aortic Stenosis; Hemodynamics
Keywords: Aortic Stenosis; Heart Valve Prosthesis; Hemodynamics; Sutureless; Standard aortic valve prosthesis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Block randomisation 1:1 of conventional Vs sutureless aortic bioprostheses.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sutureless Aortic Valve Prosthesis (Experimental): Patients receiving sutureless aortic valve prostheses
  Interventions: Device: Sutureless aortic bioprosthesis
- Conventional Aortic Valve Prosthesis (Active Comparator): Patients receiving conventional biological aortic prostheses
  Interventions: Device: Conventional stented sutured aortic prosthesis

INTERVENTIONS:
Device: Sutureless aortic bioprosthesis — Patients will receive a sutureless aortic bioprosthesis
  Arms: Sutureless Aortic Valve Prosthesis
Device: Conventional stented sutured aortic prosthesis — Patients will receive a stented sutured aortic prosthesis
  Arms: Conventional Aortic Valve Prosthesis

SUMMARY:
Multicenter randomised study which aims to compare sutureless Vs. standard bio- prostheses (1:1) among patients undergoing surgical aortic valve replacement in terms of:

* 6 -month hemodynamic performance.
* 6 month clinical outcomes including all cause mortality, stroke, myocardial infarction, valve reoperation and major/life threatening bleeding
* Cost effectiveness

DETAILED DESCRIPTION:
This study is aimed to compare clinical and hemodynamic performance of conventional sutured stented bio-prostheses among patients undergoing a surgical aortic valve replacement. The prostheses are not pre specified to be provided by a specific manufacturer, so that any bio prosthesis but transcatheter and scentless aortic valves can be implanted.

The estimated sample size is 350 patients. They will be randomised 1:1 to any of the two arms of the study (standard Vs. sutureless prostheses). The randomisation will be stratified according to the need for a concomitant coronary artery bypass grafting procedure.

Six hospitals in Madrid (Spain) will take part in the study. The period of recruitment will start as soon as June 2019 and is supposed to finish by June 2020 or earlier.

The main outcomes of the study will be measured 6 months after the aortic valve implantation

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18
* Pure aortic stenosis or combined aortic stenosis/regurgitation
* Aortic annulus >18 mm and < 27 mm

Exclusion Criteria:

* Pregnancy
* Willing to receive some other prosthesis
* Concomitant surgery of the ascending aorta or left ventricle outflow tract
* Endocarditis
* Emergency
* Some other concomitant procedure
* Participation in any other study
* Previous surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2019-06-02 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Differences in mid term trans prosthetic gradients | 6 month
  The differences in mid term trans prosthetic gradients measured by trans thoracic echocardiogram 6 months after the procedure

SECONDARY OUTCOMES:
Survival from Combined major adverse cardiovascular event | 6 month
  Comparison of survival free from a combined event including: all cause mortality, major stroke (mRS>1), Myocardial Infarction (according to VARC-II criteria), Valve re operation of any case, major or life-threatening bleeding (VARC 2 definition)
Differences in quality if life according to the KCCQ12 questionnaire | 6 month
  Quality of life will be compared between the two groups using the Kansas City Cardiomyopathy Questionnaire (KCCQ12). The response options of the items are Likert scales of 1 to 5, 6 or 7 points and the score has a theoretical range of 0 to 100, with 100 being the best

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Carnero, MD, PhD, Principal Investigator — Hospital Clinico San Carlos. Madrid. Spain
Locations (1):
- Hospital Clínico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No